CLINICAL TRIAL: NCT04177901
Title: The Use of NIRS of Monitorization in Arteriovenous Fistule Surgery With Brachial Plexus Block or Local Infiltration Anesthesia
Brief Title: The Use of NIRS in Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Tugce Topcam, doctor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0260
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Arterio-venous Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brachial plexus blockage group (Active Comparator)
  Interventions: Device: Near infrared spectroscopy
- local anesthesia group (Active Comparator)
  Interventions: Device: Near infrared spectroscopy

INTERVENTIONS:
Device: Near infrared spectroscopy — It is used for detection of tissue oxygenation

SUMMARY:
The study is planed on ASA I-III, 18-80 years old 60 patients developing chronic renal failure and needing arteriovenous fistula surgery for dialysis program in Istanbul Medeniyet University Goztepe Research Hospital. Informed consent of the patients will be obtained before surgery.Patients with hemoglobinopathy, coagulopathy, wound or infection in the thenar eminence, wound and infection in the supraclavicular region on the side of the regional block, allergic to local anesthetic drugs and mental retardation will not be included in the study.

Standart monitorization (ECG, peripheral oxygen saturation and non-invasive arterial pressure monitoring) will be made. Base and 5 minutes interval values will be recorded until the end of the surgery. The pads of the NIRS monitor will be placed on the thenar eminence of both hands and fixed with the help of a draipe and basal measurements will be taken and recorded. The patients will then be divided into two groups according to computer-generated table of random numbers.

Group L patients will undergo surgical cleansing and sterile draping and infiltrate %5 bupivacaine 15ml. Group B the supraclavicular areas of the patients who will undergo surgical procedures will be sterile covered after appropriate sterilization. After the brachial plexus is visualized around the subclavian artery in the supraclavicular region with the help of Samsung ultrasound device, Bupivacaine 5% 20ml and Lidocaine 2% 10ml will be applied around the brachial plexus using a 50mm stimuplex needle. The effectiveness of the block will be evaluated by a single investigator after withdrawal of the needle, either by effective anesthesia with the block or every 10 minutes up to 30 minutes. The sensory block will be evaluated with a 3 point scale and the motor block will be evaluated routinely before and after the modified bromage scale (scored between 0 and 4). After withdrawal of the treated needle, we will contact the relevant nerve dermatome with cold application (cold SF) and ask the patient to classify the degree of cold feeling from 0 to 3. Block will be considered unsuccessful if surgical block cannot be provided after 30 minutes or if the patient experiences pain at any time during the operation. The duration of anesthesia occurring after local infiltration of Group L and the sensory and motor blockade after group B stimulation is taken will be recorded. In both groups, NIRS values will be recorded at 5 minute intervals until the end of the case after local anesthetic application.

Investigator will call the patients for primer patency of fistula one month after operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III,
* chronic renal failure and needing arteriovenous fistula surgery

Exclusion Criteria:

* hemoglobinopathy
* coagulopathy,
* wound or infection in the thenar eminence
* wound and infection in the supraclavicular region on the side of the regional block
* allergic to local anesthetic drugs
* mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
improvement of tissue oxygenation | 85 minutes
  Improvemen of tissue oxygenation by different anesthetic technique

SECONDARY OUTCOMES:
primary patency of arteriovenous fistula | 1 month
  Patients will called after one month later from surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided